CLINICAL TRIAL: NCT01127048
Title: Investigation on Efficacy and Tolerability of Prospan® Hustenzäpfchen for the Symptomatic Treatment of Acute Bronchitis Accompanied by Coughing in Children
Brief Title: Prospan® Hustenzäpfchen - Investigation on Efficacy and Tolerability in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Engelhard Arzneimittel GmbH & Co.KG (Industry)
Responsible Party: Prof. Dr. Gerhard Zwacka, Robert-Koch-Krankenhaus Apolda
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EA-08-1-34
Record Dates: First submitted 2010-05-03; First posted 2010-05-20 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2010-05

CONDITIONS: Symptoms of Acute Bronchitis Accompanied by Coughing
Keywords: bronchitis; coughing; children; Ivy; Hedera helix L.
MeSH Terms: conditions — Bronchitis; Cough

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prospan Hustenzäpfchen (Experimental)
  Interventions: Drug: Suppositories containing Ivy leaves dry extract
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Suppositories containing Ivy leaves dry extract — Suppositories containing Ivy leaves dry extract
  Other Names: Prospan® Hustenzäpfchen
  Arms: Prospan Hustenzäpfchen
Drug: Placebo — Suppositories containing no Ivy leaves dry extract
  Arms: Placebo

SUMMARY:
The aims of this study are

* Demonstrating superior efficacy of Prospan® Hustenzäpfchen compared to Placebo in children suffering from acute bronchitis accompanied by coughing
* Characterisation of safety and tolerability of Prospan® Hustenzäpfchen in comparison with placebo.

DETAILED DESCRIPTION:
After interim analysis of the first part the clinical study will be continued as follows: Double blind, placebo controlled, randomised, multi-centre study with 2-parallel groups for the treatment of acute bronchitis accompanied by coughing in children aged 0 - 6 years to demonstrate efficacy and safety of Prospan® Hustenzäpfchen.

For assessment of cough intensity and severity a specific symptom score has been developed, which gathers the child's frequency and severity of coughing and of cough productivity as well as the severity of rhonchi (each symptom will be assessed on a four-point Likert scale ranging from 0 to 3; total score range: 0-12 points).

Considering the specificities of the study population and the disease, confirmatory evaluation will be based on the change in the symptom score after the first three consecutive days of treatment as assessed by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. male or female children aged 0 to 6 years
2. acute bronchitis existing not longer than three days and accompanied by coughing
3. symptom rating score of ≥ 5 assessed by the investigator
4. symptom 'frequency of coughing' of ≥ 2 assessed by the investigator
5. the patient's legal representatives must give informed consent in accordance with the supposed will of the patient, after having been informed about benefits and potential risks of the trial, as well as details of the insurance taken out to cover the risk for patients participating in the study -

Exclusion Criteria:

1. hypersensitivity to the active ingredient or to any further constituents of the pharmaceutical preparations
2. patients with severe allergies or multiple drug allergies
3. any other pulmonary disease within the last two weeks
4. chronic pulmonary diseases
5. exacerbation of chronic pulmonary disease
6. suspicion of bacterial pulmonary infection
7. fever above 39°C (rectal measurement) -

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1400 (Estimated)
Dates: Start 2008-10; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure | 7 days
  Effect of treatment as primary variable will be assessed by comparing baseline values to those obtained during visit 2.
  The primary outcome measure for efficacy will be the relative change in the symptom score between visits 1 and 2.

SECONDARY OUTCOMES:
Secondary variables | 7 days
  * absolute change of total symptom score
  * time to response
  * compliance, defined by drug accountability
  * percentage of patients requiring concomitant medication for treatment of cough
  * rates of premature withdrawal
  * incidence of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Zwacka, Prof. Dr., Principal Investigator
Locations (1):
- Engelhard Arzneimittel GmbH & Co. KG, Niederdorfelden, Germany